CLINICAL TRIAL: NCT01281215
Title: Education Interventions Model for Rational Drug Use
Brief Title: Education Interventions Model for Rational Drug Use (RDU)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Carolina Maria Xaubet Olivera, Masters, University of Sao Paulo
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FR - 381298
Record Dates: First submitted 2011-01-19; First posted 2011-01-21 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Asthma
Keywords: Pharmaceutical Education; Rational Drug Use; Asthma
MeSH Terms: conditions — Asthma | interventions — Pharmaceutical Services

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pharmaceutical Education (Experimental): The patients will receive pharmaceutical education.
  Interventions: Behavioral: Education interventional
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Education interventional — The patients will receive pharmaceutical education to know more about asthma, the importance of treatment compliance, the medications used to control the pathology, corrected patients' inhalation techniques and the medication care.
  Other Names: Pharmaceutical Care
  Arms: Pharmaceutical Education

SUMMARY:
The purpose of this study is to develop, implement and evaluate an economically viable and efficient interventions education model for rational drug use, adaptable to different pathological situations and should be implemented into Brazil Heath Care System.

DETAILED DESCRIPTION:
Currently, the educational interventions regarding the use of medicines need to be expanded and more effective, and thus set themselves up in strategies for reorganization of dispensing drugs in health services and provide support to the population to obtain greater control over their health. The pharmacist, in turn, inserted in the multidisciplinary team has an important role in health education with the aim of improving knowledge about the disease and the various treatment options, reflecting positively on treatment adherence and clinical outcomes as a result and quality of life related to patient health. Thus, health education, to share knowledge, represents an important task and involves attentive listening to the community to identify their needs and then solve them. From this perspective, therefore, the educational means to educate health and an integral formation of individuals as social actors critics who understand and question the social relations, transforming subjects into citizens participating in the process of health education, helping to raise awareness , knowledge and understanding of living conditions and relationships with health, promoting quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Subject with asthma diagnosed according to criteria of the Global Strategy for Asthma Management and Prevention;
* Subject is a male or female with 18 to 73 years-old;
* Subject who has access to medications supplied by the the Brazil Heath Care System;
* Subject unable to perform the procedures or conditions such as pregnancy that may affect the results of the study;
* Literate subject without Cognitive Disorders, Alzheimer's, Dementia, that can limit the ability to participate in this study;
* Subject who have availability to attend the monthly meetings;
* Subject provides written informed consent and attend the first evaluation.

Exclusion Criteria:

* Subject who cannot be classified in the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Knowledge of Asthma | 6 months after the first evaluation
  To compare the patient´s knowledge of asthma before and after the education interventions with asthma knowledge questionnaire.

SECONDARY OUTCOMES:
Spirometry Exam | 6 months after the first evaluation
  To compare the patient´s pulmonary function before and after the education interventions with spirometry exam.
Sociodemographic data, clinical and lifestyle evaluation | 6 months after the first evaluation
  To evaluate the sociodemographic data, clinical and lifestyle before and after the education interventions and its impact on the quality of life.
Management of inhalers | 6 months after the first evaluation
  To evaluate the technique for using inhalation devices among asthma patients before and after education interventions. Patients will be asked to demonstrate their inhaler technique.
Treatment compliance evaluation | 6 months after the first evaluation
  To evaluate the treatment compliance with Morisky&Green test and pharmacy database query before and after educations interventions.
Economic analysis | 6 months after the first evaluation
  Economic analysis after the model implementation.
Quality of Life Evaluation | 6 months after the first evaluation
  To compare the Quality of Life before and after the education interventions

CONTACTS AND LOCATIONS:
Overall Officials: Osvaldo de Freitas, habilitation, Study Director — Pharmaceutical Sciences Faculty of Ribeirão Preto, University of São Paolo; Elcio Vianna, habilitation, Study Director — Clinical Hospital of Medicine Faculty of Ribeirão Preto, University of São Paolo; Carolina Olivera, Masters, Principal Investigator — Pharmaceutical Sciences Faculty of Ribeirão Preto, University of São Paolo
Locations (1):
- Clinical Hospital of Medicine Faculty of Ribeirão Preto, University of São Paolo, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Derived] Olivera CM, Vianna EO, Bonizio RC, de Menezes MB, Ferraz E, Cetlin AA, Valdevite LM, Almeida GA, Araujo AS, Simoneti CS, de Freitas A, Lizzi EA, Borges MC, de Freitas O. Asthma self-management model: randomized controlled trial. Health Educ Res. 2016 Oct;31(5):639-52. doi: 10.1093/her/cyw035. Epub 2016 Jul 29. PMID 27473571